CLINICAL TRIAL: NCT04821492
Title: Evaluation of the Relationship Between Homocysteine Levels and Bone Mineral Density in Postmenopausal Women
Brief Title: Relationship Between Homocysteine and BMD
Status: Completed | Type: Observational
Sponsor: Fundación Santiago Dexeus Font (Other)
Responsible Party: Principal Investigator, Pascual García, Principal Investigator, Fundacion Dexeus
Organization: Fundacion Dexeus (Other)
Other Study IDs: FSD-HCY-2020-05
Record Dates: First submitted 2021-03-24; First posted 2021-03-29 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2021-03

CONDITIONS: Postmenopausal Women
MeSH Terms: interventions — Absorptiometry, Photon

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hyperhomocysteinemia
  Interventions: Diagnostic Test: Dual-Energy X-ray Absorptiometry (DXA)
- Normal Hcy levels
  Interventions: Diagnostic Test: Dual-Energy X-ray Absorptiometry (DXA)

INTERVENTIONS:
Diagnostic Test: Dual-Energy X-ray Absorptiometry (DXA) — BMD expressed in absolute values as g/cm2 and T-scores

SUMMARY:
The association between Homocysteine (Hcy) levels and bone mineral density (BMD) has been debated. Some studies have found a relationship between increased Hcy plasma levels and BMD in contrast; other studies have not found a relationship. The purpose of our study was to investigate whether or not Hcy plasma levels are related to BMD in a group of postmenopausal women.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women
* BMD measured by dual-energy X-ray absorptiometry (DXA)

Exclusion Criteria:

* Primary ovarian failure
* Early menopause
* Cardiovascular, liver, or renal diseases
* Surgical menopause
* History of cancer
* Receiving treatment known to influence levels of Hcy or bone mineralization (folates or vitamin B12 supplements, menopausal hormonal treatment, corticosteroids, anticonvulsants, heparin, thiazide diuretics, and antiresorptive agents).

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women visited at the Obstetrics and Gynecology Department at the Hospital Universitario Dexeus (Barcelona, Spain).
Sampling Method: Non-Probability Sample
Enrollment: 760 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
BMD expressed in absolute values as g/cm2 | one year before or after Homocysteine levels
Lumbar spine T-score | one year before or after Homocysteine levels
Femoral neck T-score | one year before or after Homocysteine levels
Total hip T-score | one year before or after Homocysteine levels

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Quiron Dexeus, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cagnacci A, Bagni B, Zini A, Cannoletta M, Generali M, Volpe A. Relation of folates, vitamin B12 and homocysteine to vertebral bone mineral density change in postmenopausal women. A five-year longitudinal evaluation. Bone. 2008 Feb;42(2):314-20. doi: 10.1016/j.bone.2007.10.022. Epub 2007 Nov 12. PMID 18289506
- [Background] Mittal M, Verma R, Mishra A, Singh A, Kumar V, Sawlani KK, Ahmad MK, Mishra P, Gaur R. Relation of Bone Mineral Density with Homocysteine and Cathepsin K levels in Postmenopausal Women. Indian J Endocrinol Metab. 2018 Mar-Apr;22(2):261-266. doi: 10.4103/ijem.IJEM_575_17. PMID 29911042
- [Background] Enneman AW, Swart KM, Zillikens MC, van Dijk SC, van Wijngaarden JP, Brouwer-Brolsma EM, Dhonukshe-Rutten RA, Hofman A, Rivadeneira F, van der Cammen TJ, Lips P, de Groot CP, Uitterlinden AG, van Meurs JB, van Schoor NM, van der Velde N. The association between plasma homocysteine levels and bone quality and bone mineral density parameters in older persons. Bone. 2014 Jun;63:141-6. doi: 10.1016/j.bone.2014.03.002. Epub 2014 Mar 12. PMID 24631997
- [Background] Bahtiri E, Islami H, Rexhepi S, Qorraj-Bytyqi H, Thaci K, Thaci S, Karakulak C, Hoxha R. Relationship of homocysteine levels with lumbar spine and femur neck BMD in postmenopausal women. Acta Reumatol Port. 2015 Oct-Dec;40(4):355-62. PMID 26922199
- See also: Related Info — http://dexeus.com